CLINICAL TRIAL: NCT02644694
Title: A Prospective, Multi-Center, Single-Dose, Phase 1 Clinical Trial Designed to Evaluate the Pharmacokinetics of Dexamethasone Phosphate Ophthalmic Solution Delivered Via the EyeGate® II Drug Delivery System in Patients Undergoing Vitrectomy for Macular Hole Repair or Epiretinal Membrane Peeling
Brief Title: PK Study of Iontophoretic Dexamethasone Phosphate Ophthalmic Solution in Patients Undergoing Vitrectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGP-437-010
Record Dates: First submitted 2015-12-22; First posted 2016-01-01 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-06

CONDITIONS: Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexamethasone Phosphate Ophthalmic Solution (Experimental): Experimental: Dexamethasone Phosphate Ophthalmic Solution (40 mg/mL) delivered via the EyeGate II Drug Delivery System
  Interventions: Drug: Dexamethasone Phosphate Ophthalmic Solution

INTERVENTIONS:
Drug: Dexamethasone Phosphate Ophthalmic Solution — Experimental: Dexamethasone Phosphate Ophthalmic Solution (40 mg/mL) delivered via the EyeGate II Drug Delivery System

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of dexamethasone phosphate ophthalmic solution delivered via the EyeGate® II Drug Delivery System (EGDS) in patients undergoing vitrectomy for macular hole repair or epiretinal membrane peeling

DETAILED DESCRIPTION:
This is an open-label, multi-center, single-dose, Phase 1 clinical trial designed to evaluate the pharmacokinetics (PK) of dexamethasone phosphate ophthalmic solution delivered via the EyeGate® II Drug Delivery System (EGDS) in the vitreous humor taken from patients undergoing vitrectomy for macular hole repair or epiretinal membrane peeling

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years
2. Receive, understand, and sign a copy of the written informed consent form

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Concentration of dexamethasone | Day 1
  Vitreous humor samples will be analyzed for dexamethasone concentrations
Concentration of dexamethasone phosphate | Day 1
  Vitreous humor samples will be analyzed for dexamethasone phosphate concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Heier, M.D., Principal Investigator — Study Principal Investigator
Locations (1):
- Ophthalmic Consultants of Boston, Boston, Massachusetts, United States